CLINICAL TRIAL: NCT00289705
Title: Surgical Intervention With Laparoscopic Roux-en-Y Gastric Bypass for Morbid Obesity in Adolescence - a Matched Control Study
Brief Title: Surgical Intervention for Morbidly Obese Adolescents
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SU523-04
Record Dates: First submitted 2006-02-09; First posted 2006-02-10 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-02

CONDITIONS: Obesity; Diabetes; Hypertension
Keywords: Obesity; Surgery; Adolescent; Roux-en-Y gastric bypass; Laparoscopic
MeSH Terms: conditions — Obesity; Diabetes Mellitus; Hypertension | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Surgery (Experimental): Laparoscopic gastric bypass
  Interventions: Procedure: Surgery
- 2 (No Intervention): Traditional treatment for obesity

INTERVENTIONS:
Procedure: Surgery — Laparoscopic Roux-en-Y gastric bypass
  Arms: Surgery

SUMMARY:
The purpose is to study whether the positive effects from obesity surgery in adults also can be achieved when adolescent subjects are operated.

Our hypothesis is that the effects concerning weight loss, health improvement and improved quality of life will be as good in adolescents as in adults.

DETAILED DESCRIPTION:
Severe obesity in the adolescence is a major concern since there is a constant rise in prevalence worldwide. There is a need of effective tools to treat those patients since the natural course with conservative treatment is very pessimistic. I. e. most of the subjects having a BMI >40kg/m2 in the adolescence will remain morbidly obese also in their adult life.

The three largest centres in Sweden treating obese children (Stockholm, Gothenburg and Malmö) will offer patients fulfilling the inclusion criteria to be operated with laparoscopic gastric bypass. If not willing to be operated they could join the study as a control case.

Subjects will be investigated at the baseline concerning physical health status and existence of medical risk factors but also regarding their quality of life, eating habits and physical activity. They will subsequently be follow over a ten year period regarding these variables.

ELIGIBILITY:
Inclusion Criteria:

* BMI >40 kg/m2 or BMI>35 with comorbidity
* Pass psychological evaluation
* Puberty status Tanner 4-5
* At least one year with active conservative treatment that failed

Exclusion Criteria:

* Lack of compliance
* Specific obesity syndrome as Praeder Willis
* Obesity due to brain injury
* Severe general disease
* Specific genetic defect (MC4R, Leptin deficiency)

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2006-02; Primary Completion 2017-11 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
BMI development | 10 years

SECONDARY OUTCOMES:
Medical risk factors, incidence of diseases (such as diabetes, hypertension etc), quality of life, socioeconomic development, eating pattern. | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Torsten Olbers, MD, PhD, Principal Investigator — Sahlgrenska University Hospital; Clude Marcus, Prof, MD, Study Chair — Dept of Pediatrics, Karolinska University Hospital, Huddinge; Staffan Mårild, MD, PhD, Study Chair — Queen Silvias Childs Hospital, Gothenburg; Carl-Erik Flodmark, MD, PhD, Study Chair — Dept of Pediatrics, MAS, Malmö
Locations (4):
- Sweden (4):
  - Sahlgrenska University Hospital, Dept of Surgery, Gothenburg, Gothenburg
  - Queen Silvias Children Hospital, Gothenburg, Göteborg
  - Dept of Pediatrics, MAS, Malmo, Malmö
  - National center for child obesity, Karolinska Huddinge, Stockholm, Stockholm County

REFERENCES:
- [Derived] Jarvholm K, Olbers T, Peltonen M, Marcus C, Flodmark CE, Gronowitz E, Dahlgren J, Karlsson J. Depression, anxiety, and suicidal ideation in young adults 5 years after undergoing bariatric surgery as adolescents. Eat Weight Disord. 2021 May;26(4):1211-1221. doi: 10.1007/s40519-020-01024-0. Epub 2020 Oct 20. PMID 33079376
- [Derived] Jarvholm K, Bruze G, Peltonen M, Marcus C, Flodmark CE, Henfridsson P, Beamish AJ, Gronowitz E, Dahlgren J, Karlsson J, Olbers T. 5-year mental health and eating pattern outcomes following bariatric surgery in adolescents: a prospective cohort study. Lancet Child Adolesc Health. 2020 Mar;4(3):210-219. doi: 10.1016/S2352-4642(20)30024-9. Epub 2020 Jan 21. PMID 31978372
- [Derived] Olbers T, Beamish AJ, Gronowitz E, Flodmark CE, Dahlgren J, Bruze G, Ekbom K, Friberg P, Gothberg G, Jarvholm K, Karlsson J, Marild S, Neovius M, Peltonen M, Marcus C. Laparoscopic Roux-en-Y gastric bypass in adolescents with severe obesity (AMOS): a prospective, 5-year, Swedish nationwide study. Lancet Diabetes Endocrinol. 2017 Mar;5(3):174-183. doi: 10.1016/S2213-8587(16)30424-7. Epub 2017 Jan 6. PMID 28065734
- [Derived] Beamish AJ, Gronowitz E, Olbers T, Flodmark CE, Marcus C, Dahlgren J. Body composition and bone health in adolescents after Roux-en-Y gastric bypass for severe obesity. Pediatr Obes. 2017 Jun;12(3):239-246. doi: 10.1111/ijpo.12134. Epub 2016 Apr 12. PMID 27071497
- [Derived] Gothberg G, Gronowitz E, Flodmark CE, Dahlgren J, Ekbom K, Marild S, Marcus C, Olbers T. Laparoscopic Roux-en-Y gastric bypass in adolescents with morbid obesity--surgical aspects and clinical outcome. Semin Pediatr Surg. 2014 Feb;23(1):11-6. doi: 10.1053/j.sempedsurg.2013.10.015. Epub 2013 Nov 15. PMID 24491362